CLINICAL TRIAL: NCT05685940
Title: Evaluation of the Predictive Value of Early Serum Trough Concentrations and Anti-drug Antibodies of Risankizumab and the Development of a Response-concentration Curve for Risankizumab in Patients With Psoriasis
Brief Title: Therapeutic Drug Monitoring of Risankizumab in Psoriasis Patients (BIOLOPTIM-RIS)
Acronym: BIOLOPTIM-RIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOLOPTIM-RIS
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Psoriasis Vulgaris
Keywords: Therapeutic drug monitoring; Psoriasis; Risankizumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: A prospective, open label, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care - risankizumab (Experimental): Patients will continue to receive risankizumab according to the standard dosing schedule: subcutaneous injections at weeks 0 and 4, then every 12 weeks (2x 75mg).
  Interventions: Procedure: Venapuncture; Procedure: Patient questionnaires

INTERVENTIONS:
Procedure: Venapuncture — Blood samples will be collected to determine the serum trough levels and anti-drug antibodies of risankizumab.
Procedure: Patient questionnaires — The study participants will complete the Dermatology Quality of Life (DLQI) and EQ-5D-5L questionnaire at each study visit.

SUMMARY:
Biologics such as risankizumab are currently the most effective treatment option for patients with moderate to severe psoriasis. But they are costly for healthcare systems and still described according to a 'one dose fits all' dosing regimen, leading to potential over-and undertreatment. In this study the investigators aim to investigate the predictive value of early serum trough levels of risankizumab and determine the therapeutic window of risankizumab in psoriasis patients.

DETAILED DESCRIPTION:
Patients will be included after signing informed consent. After inclusion, patients will continue on standard dosing schedule of risankizumab (i.e. subcutaneous injections at weeks 0 and 4, then every 12 weeks (2x 75mg)). During each study visit blood will be taken in order to quantify Ctroughs and/or anti-drug antibodies towards risankizumab. In addition, Psoriasis Area and Severity Index (PASI) and Investigator's Global Assessment (IGA) score will be evaluated by a physician. Patients complete the Dermatology Life Quality Index (DLQI) and European quality of life EQ-5D instrument at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a clinical or histological diagnosis of chronic plaque-type psoriasis
* Participants must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Exclusion Criteria:

* Participants who have currently a predominant nonplaque form of psoriasis
* Participants who are pregnant, nursing or planning a pregnancy
* Participants who are unable or unwilling to undergo multiple venapunctures
* Participants who are treated according to a different dosing schedule than standard dosing of risankizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of early serum trough concentrations of risankizumab | Week 0 until week 24 of treatment
  To assess the predictive value of early serum trough levels of risankizumab (µg/ml), the clinical response (PASI) at week 12 and/or week 24 will be correlated with serum trough concentrations of tildrakizumab measurements taken from week 0,1,2,3 and/or 4.
Predictive value of early anti-drug antibodies of risankizumab | Week 0 until week 24 of treatment
  To assess the predictive value of early anti-drug antibodies of risankizumab (µg/ml), the clinical response (PASI) at week 12 and/or week 24 will be correlated with anti-drug antibodies of tildrakizumab measurements taken from week 0,1,2,3 and/or 4.
Development of the therapeutic window of risankizumab in psoriasis | Week 0 until week 52 of treatment
  Defining a therapeutic window for risankizumab based on serum trough concentrations corresponding with adequate clinical response (ROC analysis and concentration-effect curve)

SECONDARY OUTCOMES:
DLQI | Week 0 until week 52 of treatment
  The DLQI (Dermatology Life Quality Index) (range 0-30) is a dermatology specific quality of life (QoL) instrument designed to assess the impact of the disease on participant's QoL. It is a ten item questionnaire that, in addition to evaluated overall QoL, can be used to assess six different aspects that may affect QoL: 1) symptoms and feelings, 2) daily activities, 3) leasure, 4) work or school performances, 5) personal relationships, and 6) treatment.
  The scoring of each question is as follows:
  Very much - scored 3; A lot - scored 2; A little - scored 1; Not at all - scored 0; Not relevant - scored 0; Question 7, 'prevented work or studying' - scored 3. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
EQ-5D-5L | Week 0 until week 52 of treatment
  The EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits of the five dimensions can be combined into a 5- digit number that describes the patients' health state.
EQ VAS | Week 0 until week 52 of treatment
  The EQ VAS (Visual Analogue Scale) (range 0-10) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof., Principal Investigator — University Ghent
Locations (7):
- Belgium (7):
  - AZ Maria Middelares, Ghent, East-Flanders
  - AZ Sint-Lucas, Ghent, East-Flanders
  - University Hospital Ghent, Ghent, East-Flanders
  - Private practice Dermatology, Maldegem, East-Flanders
  - University Hospital Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan, Bruges, West-Flanders
  - AZ Delta Rembert, Torhout, West-Flanders

IPD SHARING:
Plan to Share IPD: No